CLINICAL TRIAL: NCT01278927
Title: A Phase III Randomized, Multicenter Trial Testing Whether Exercise or Stress Management Improves Functional Status and Symptoms of Autologous and Allogeneic Recipients (BMT CTN #0902)
Brief Title: Exercise and Stress Management Post Autologous and Allogeneic Transplant (BMT CTN 0902)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: BMTCTN0902; U01HL069294 (NIH); BMT CTN 0902 (Other: Blood and Marrow Transplant Center Clinical Trials Network); 5U24CA076518 (NIH)
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Physiological Stress
Keywords: exercise; stress management; post transplant; physical and emotional relaxation
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Restraint, Physical; Standard of Care; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Exercise (Active Comparator): Participants assigned to the Exercise arm will receive a packet of materials from the study interventionist, along with a brief (10 minute) personalized introduction to the home-based exercise intervention. On Day 30 post hematopoietic cell transplantation (HCT), participants will meet briefly with the same interventionist when possible. To minimize contamination across intervention conditions, participants randomized to Exercise will be provided with only general advice regarding stress management (i.e., to continue using any techniques they currently use to manage stress). The interventionist will meet with the patient again in person or by phone at approximately 60 days post transplant.
  Interventions: Behavioral: Exercise
- Stress Management (Active Comparator): Participants will receive a packet of materials from the study interventionist, along with a brief standardized introduction to the self-administered intervention. On Day 30 post HCT, the interventionist will meet with the participant to answer any questions about the intervention, encourage the continued use of stress management techniques as recommended, and monitor for any adverse reactions to use of the techniques. The interventionist will meet with the patient again in person or by phone at approximately 60 days post transplant. Whenever possible, the interventionist meeting with the patient at 30 and 60 days should be the same interventionist who previously met with the patient.
  Interventions: Behavioral: Stress Management
- Exercise and Stress Management (Active Comparator): Participants will receive a packet of materials from the study interventionist, along with a brief (15 minute) personalized introduction to the interventions. On Day 30 post HCT, the same interventionist will meet with the participant briefly to answer any questions about the interventions, encourage the continued use of the interventions as recommended, and monitor for any adverse reactions. The interventionist will meet with the patient again in person or by phone at approximately 60 days post transplant. Whenever possible, the interventionist meeting with the patient at 30 and 60 days should be the same interventionist who previously met with the patient.
  Interventions: Behavioral: Exercise and Stress Management
- Standard Care (Other): Patients randomized to standard care only will be informed of their assigned condition and receive a digital video disc (DVD). The interventionist will briefly discuss the topics of the DVD and elicit questions. To minimize contamination across intervention conditions, participants randomized to the control group will be provided with only general advice about exercise and stress management during treatment (i.e., to maintain any usual patterns of exercise to the extent possible and to continue using any techniques they currently use to manage stress).
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Exercise — Participants assigned to the Exercise arm will receive a packet of materials from the study interventionist, along with a brief personalized introduction to the home-based exercise intervention.
  Other Names: Physical activities; Musculoskeletal; Exertian level
  Arms: Exercise
Behavioral: Stress Management — Participants will receive a packet of materials from the study interventionist, along with a brief (10 minute) standardized introduction to the self-administered intervention.
  Other Names: Active relaxation; Deep breathing; Positive thinking; Relaxing
  Arms: Stress Management
Behavioral: Exercise and Stress Management — Participants will receive a packet of materials from the study interventionist, along with a brief (15 minute) personalized introduction to the interventions.
  Other Names: Physical and emotional relaxation; Active relaxation
  Arms: Exercise and Stress Management
Other: Standard Care — Patients randomized to standard care only will be informed of their assigned condition and receive the DVD.
  Other Names: General care; Psychosocial care
  Arms: Standard Care

SUMMARY:
This is a Phase III, randomized, unblinded, multicenter, prospective comparative study. The purpose of this study is to test whether exercise or stress management training delivered to autologous and allogeneic hematopoietic cell transplantation (HCT) patients prior to transplantation can improve functional status and the transplant experience.

DETAILED DESCRIPTION:
Background:

The adverse effects of hematopoietic cell transplantation (HCT) on short and long term quality of life are well documented. Patients experience numerous aversive symptoms (e.g., nausea, fatigue, and sleep disturbance) that are accompanied by declines in physical and mental well-being. Although most longitudinal studies show return to baseline functioning for the majority of patients, it may take 6 to 12 months or longer to reach this goal. Clinical trials have shown that training in stress management techniques and participation in formal exercise programs each offered in isolation are effective in improving quality of life in patients receiving standard-dose chemotherapy and HCT. Review of these studies suggests that stress management interventions primarily improve mental health outcomes and nausea. The impact of exercise training interventions is more variable; most studies report physical health benefits, with some studies also reporting mental health benefits. Small studies suggest that combining stress management training and exercise are feasible and well-tolerated, but whether the combination provides an additive or synergistic impact on quality of life outcomes has not been directly investigated.

Design Narrative:

The protocol is designed as a factorial trial with two interventions, exercise and stress management, which results in four treatment arms: standard care, exercise only, stress management only and the combination of exercise and stress management. The primary objective of this randomized phase III trial is to test the ability of exercise training or stress management training to improve physical and mental functioning at Day 100 post hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to speak and read English
* Able to exercise at low to moderate intensity - adequate cardiopulmonary reserve, as judged by self-reported ability to walk up one flight of stairs, no requirement for supplemental oxygen, and physician judgment
* Willing and able to provide informed consent.
* Stated willingness to comply with study procedures and reporting requirements
* Planned autologous or allogeneic transplantation within 6 weeks.

Exclusion Criteria:

* Orthopedic, neurologic or other problems which prevent safe ambulation and protocol adherence
* Participation in another clinical trial with quality of life or functional status as a primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (19):
- United States (19):
  - City of Hope National Medical Center, Duarte, California
  - University of Florida College of Medicine, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Blood & Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase, Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - Virginia Commonwealth University, MCV Hospital, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Jacobsen PB, Le-Rademacher J, Jim H, Syrjala K, Wingard JR, Logan B, Wu J, Majhail NS, Wood W, Rizzo JD, Geller NL, Kitko C, Faber E, Abidi MH, Slater S, Horowitz MM, Lee SJ. Exercise and stress management training prior to hematopoietic cell transplantation: Blood and Marrow Transplant Clinical Trials Network (BMT CTN) 0902. Biol Blood Marrow Transplant. 2014 Oct;20(10):1530-6. doi: 10.1016/j.bbmt.2014.05.027. Epub 2014 Jun 6. PMID 24910380
- [Result] Wood WA, Le-Rademacher J, Syrjala KL, Jim H, Jacobsen PB, Knight JM, Abidi MH, Wingard JR, Majhail NS, Geller NL, Rizzo JD, Fei M, Wu J, Horowitz MM, Lee SJ. Patient-reported physical functioning predicts the success of hematopoietic cell transplantation (BMT CTN 0902). Cancer. 2016 Jan 1;122(1):91-8. doi: 10.1002/cncr.29717. Epub 2015 Oct 6. PMID 26439325

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Started | 180 | 178 | 178 | 175
Completed | 180 | 178 | 178 | 175
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care | Total
Number analyzed (Participants) | 180 | 178 | 178 | 175 | 711
Age, Customized [Number; unit: participants]
  <=40 years | 26 | 21 | 26 | 27 | 100
  41-<65 years | 105 | 123 | 118 | 111 | 457
  >=65 years | 49 | 34 | 34 | 37 | 154
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 78 | 78 | 82 | 306
  Male | 112 | 100 | 100 | 93 | 405
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 11 | 6 | 35
  Not Hispanic or Latino | 172 | 167 | 167 | 167 | 673
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 3 | 4 | 2 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 1 | 3
  Black or African American | 14 | 17 | 13 | 16 | 60
  White | 162 | 152 | 160 | 152 | 626
  More than one race | 0 | 1 | 2 | 3 | 6
  Unknown or Not Reported | 0 | 3 | 0 | 1 | 4
Karnofsky Performance-status Score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    >=90% | 112 | 111 | 94 | 102 | 419
    70%-80% | 65 | 64 | 76 | 68 | 273
    50%-60% | 2 | 1 | 3 | 4 | 10
    Missing/Not done | 1 | 2 | 5 | 1 | 9
Disease [Number; unit: participants]
  AML/ANLL/ALL | 42 | 47 | 40 | 42 | 171
  CML | 5 | 5 | 2 | 2 | 14
  MDS/MPS | 19 | 16 | 15 | 13 | 63
  MM/PCD | 50 | 44 | 45 | 57 | 196
  Lymphoma | 54 | 60 | 66 | 50 | 230
  CLL/SLL | 5 | 3 | 5 | 7 | 20
  Solid Tumors | 0 | 1 | 0 | 1 | 2
  SAA | 3 | 2 | 2 | 2 | 9
  Other Disease | 1 | 0 | 0 | 0 | 1
  Missing | 1 | 0 | 3 | 1 | 5

OUTCOME MEASURES:

1. Secondary Outcome: Symptoms
Description: Patients will complete the MOS 36-Item Short Form (SF-36), a widely used self-report measure designed to assess perceived health and functioning, contains eight scales: Physical Functioning (PF), Role-Physical (R-P); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Mental Health (MH); and Role-Emotional (R-E). Scales are comprised of different numbers of items and use a variety of rating formats. Raw scores are converted to a standard metric (0-100), with higher scores being indicative of a better health state.
Time Frame: 100 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 139 | 142 | 136 | 143
units on a scale
  Physical Functioning | 66.46 (24.47) | 66.12 (23.95) | 65.83 (23.34) | 67.38 (24.30)
  Role Physical | 54.79 (30.21) | 53.49 (30.72) | 54.74 (29.33) | 58.51 (26.98)
  Bodily Pain | 67.78 (24.74) | 71.55 (25.17) | 67.96 (26.18) | 68.19 (24.15)
  General Health | 63.62 (19.93) | 60.05 (19.86) | 58.06 (20.25) | 59.43 (19.38)
  Vitality | 54.91 (20.84) | 58.13 (18.29) | 54.42 (21.03) | 53.56 (21.06)
  Social Functioning | 73.83 (25.89) | 76.13 (26.52) | 72.64 (26.96) | 72.67 (26.68)
  Role Emotional | 81.73 (25.64) | 80.44 (26.83) | 86.68 (21.23) | 81.83 (25.29)
  Mental Health | 76.68 (17.24) | 80.17 (15.29) | 77.85 (17.58) | 76.75 (17.59)

2. Primary Outcome: Functional Status
Description: To determine whether exercise or stress management improves self-reported physical and mental functioning compared to standard care at 100 days post hematopoietic cell transplantation (HCT) using evaluated patients. The Physical Component Score (PCS) and Mental Component Score (MCS) of the SF-36 will be the primary endpoint measures of functional status. Raw scores are converted to a standard metric (0-100), with higher scores being indicative of a better health state.
Time Frame: 100 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 139 | 142 | 136 | 143
units on a scale
  PCS | 42.2 (10.47) | 41.8 (9.59) | 40.6 (10.49) | 42.5 (9.22)
  MCS | 50.8 (10.44) | 52.4 (9.43) | 52.1 (9.70) | 50.4 (10.69)

3. Secondary Outcome: Cancer and Treatment Distress (CTXD)
Description: Cancer and treatment distress will be measured by the acute version of the Cancer and Treatment Distress (CTXD) scale, a 27 item validated measure of distress with domains of Uncertainty, Health Burden, Family Strain, Identity and Managing the Medical System used extensively in HCT studies. The scale ranges from 0 - 3, where a higher score reflects more distress.
Time Frame: 100 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 140 | 144 | 138 | 144
units on a scale | 0.96 (0.56) | 0.88 (0.60) | 1.04 (0.66) | 0.94 (0.57)

4. Secondary Outcome: The Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a widely used seven item self-report measure of sleep patterns and difficulties. A modified version will be used to obtain self-reports of the following for the past week: sleep quality, sleep latency, sleep efficiency, and use of sleeping medications. The scale ranges from 0 - 21, where a higher score reflects worse sleep quality.
Time Frame: 100 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 132 | 136 | 135 | 138
units on a scale | 4.55 (3.50) | 3.49 (2.93) | 4.44 (3.31) | 4.02 (3.13)

5. Secondary Outcome: Nausea
Description: Two questions using a similar format as the SF-36 were added to measure nausea. The scale ranges from 1 - 5, where a higher score indicates worse nausea.
Time Frame: 100 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 138 | 143 | 138 | 144
units on a scale | 2.74 (1.38) | 2.63 (1.41) | 2.80 (1.47) | 2.85 (1.49)

6. Secondary Outcome: Days of Hospitalization
Description: The number of hospital days within the first 100 days after graft infusion will be collected for patients surviving at least 100 days.
Time Frame: 100 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 175 | 172 | 172 | 173
days | 21.1 (20.3) | 22.7 (19.6) | 21.6 (20.6) | 20.9 (17.0)

7. Secondary Outcome: SF-36 Late Outcomes
Description: The SF-36 PCS and MCS will be collected from participants at six months. Raw scores are converted to a standard metric (0-100), with higher scores being indicative of a better health state.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 125 | 122 | 117 | 128
units on a scale
  PCS | 44.5 (9.4) | 42.3 (10.6) | 43.4 (10.0) | 42.8 (10.1)
  MCS | 51.6 (9.8) | 52.5 (9.1) | 50.7 (11.0) | 51.7 (9.9)

8. Secondary Outcome: Survival
Description: Both survival at 6 months and overall survival at last follow-up will be reported. Overall survival is defined as the interval between transplantation and death or last follow-up. Patients alive when the study closes or lost to follow up are censored at the date of last contact.
Time Frame: 6 months and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Exercise and Stress Management: Exercise and Stress Management - Participants will receive a packet of materials from the study interventionist, along with a brief (15 minute) personalized introduction to the interventions.
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Number analyzed (Participants) | 180 | 178 | 178 | 175
percentage of participants
  6 months | 89 [83 to 92] | 89 [84 to 93] | 86 [80 to 90] | 92 [88 to 96]
  1 year | 85 [79 to 90] | 82 [75 to 88] | 72 [64 to 80] | 79 [70 to 86]

ADVERSE EVENTS:
Time Frame: 6-months post-transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event.
Arm/Group | Exercise | Stress Management | Exercise and Stress Management | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/178 | 0/175 | 1/174 | 0/174
Other Adverse Events (participants affected / at risk) | 0/178 | 0/175 | 0/174 | 0/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise (N=178) | Stress Management (N=175) | Exercise and Stress Management (N=174) | Standard Care (N=174)
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-03-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT01278927/Prot_SAP_ICF_000.pdf